CLINICAL TRIAL: NCT05058456
Title: Prospective, Multi-center, Single-arm Feasibility Study of the Shockwave Medical Mini S Peripheral Intravascular Lithotripsy (IVL) System
Brief Title: Mini S Feasibility Study With Shockwave Medical Mini S Peripheral IVL System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP 65324
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental)
  Interventions: Device: Shockwave Medical Mini S Peripheral IVL Catheter

INTERVENTIONS:
Device: Shockwave Medical Mini S Peripheral IVL Catheter — The Shockwave Medical Mini S Peripheral IVL Catheter is intended for lithotripsy-enhanced catheter dilatation of lesions, including calcified lesions found in the peripheral vasculature, such as the iliac, femoral, ilio-femoral, popliteal, infra-popliteal, and renal arteries. The Mini S IVL Catheter is not for use in the coronary or cerebral vasculature.

SUMMARY:
Prospective, multi-center, single-arm feasibility study to assess the safety and performance of the Shockwave Medical Mini S Peripheral IVL System for the treatment of heavily calcified, stenotic peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

-General Inclusion Criteria

1. Age of subject is ≥ 18 years.
2. Subject is able and willing to comply with all assessments in the study.
3. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
4. Estimated life expectancy > 1 year.
5. Rutherford Clinical Category 2, 3, 4 or 5 of the target limb(s).

   * Angiographic Inclusion Criteria
6. One or two target lesion(s) located in a native de novo superficial femoral, popliteal or infrapopliteal artery (above the ankle joint), in one or both limbs.
7. Target lesion reference vessel diameter (RVD) between 2.0 mm and 7.0 mm by investigator visual estimate.
8. Target lesion stenosis ≥70% (for vessels below the knee defined as P3 to the ankle joint) or ≥90% (for vessels above the knee) by investigator visual estimate.
9. Target lesion length is ≤150 mm by investigator visual estimate. Target lesion can be all or part of the 150 mm treated zone.
10. Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

Exclusion Criteria:

- General Exclusion Criteria

1. Rutherford Clinical Category 0, 1 and 6 (target limb).
2. History of endovascular or surgical procedure on the target limb within the last 30 days, or planned within 30 days of the index procedure. Note: inflow treatment of non-target lesions is allowed providing successful treatment.
3. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
4. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
5. Subject has known allergy to urethane, nylon, or silicone.
6. Myocardial infarction within 60 days prior to enrollment.
7. History of stroke within 60 days prior to enrollment.
8. Subject has acute or chronic renal disease with eGFR <30 ml/min/1.73 m2 (using CKD-EPI formula), unless on renal replacement therapy.
9. Subject is pregnant or nursing.
10. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
11. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
12. Covid-19 diagnosis within 30 days.
13. Planned use of cutting/scoring balloons, re-entry or atherectomy devices in target lesion(s) during the index procedure.
14. Planned major amputation of target limb.
15. Acute limb ischemia.
16. Occlusion of all the inframalleolar outflow arteries/vessels (i.e., desert foot).
17. Subject already enrolled into this study.

    * Angiographic Exclusion Criteria
18. Failure to treat clinically significant inflow lesions in the ipsilateral iliac, femoral, or popliteal arteries with ≤30% residual stenosis, and no serious angiographic complications (e.g. embolism).
19. Failure to successfully treat significant non-target infra-popliteal lesions, if treated prior to target lesion(s). Successful treatment is defined as obtaining ≤50% residual stenosis with no serious angiographic complications (e.g., embolism).
20. Target lesion includes in-stent restenosis.
21. Evidence of aneurysm or thrombus in target vessel.
22. No calcium or mild calcium in the target lesion.
23. Target lesion within native or synthetic vessel grafts.
24. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - Sir Charles Gairdner Hospital, Nedlands, Perth
  - Royal Perth Hospital, Perth
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-arm
Started | 35
30 Days Post-Procedure | 34
Completed | 0 (End of Study data not yet due for release)
Not Completed | 35
Not completed — Death | 1
Not completed — End of Study data not yet due for release | 34

BASELINE CHARACTERISTICS:
Arm/Group | Single-arm
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  New Zealand | 22
  Australia | 13

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety: Major Adverse Events (MAE)
Description: Major Adverse Events (MAE) at 30 days defined as a composite of:
  * Cardiovascular Death
  * Clinically Driven Target Lesion Revascularization (CD-TLR)
  * Unplanned Target Limb Major Amputation (Above the Ankle)
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Single-arm
Number analyzed (Participants) | 35
participants
  Major Adverse Events | 1
  Cardiovascular Death | 1
  Clinically-Driven Target Lesion Revascularization (CD-TLR) | 0
  Unplanned Target Limb Major Amputation (Above the Ankle) | 0
Statistical Analysis 1: Comparison: Single-arm; Test type: Other — The primary safety hypothesis is: H0: ΠS > PGS vs. HA: ΠS ≤ PGS where ΠS is the proportion of patients who experience a MAE within 30 days of procedure and PGS is the Safety Performance Goal. All subjects in whom a Mini S IVL catheter was introduced into the vasculature will be included in the analysis (i.e., it is an intent-to-treat analysis). The hypothesis will be tested using a one-sided Exact Binomial Test at α=0.025; p < .025, Fisher Exact

2. Primary Outcome: Primary Performance: Technical Success
Description: Technical Success defined as final residual stenosis ≤50% without flow-limiting dissection (≥ Grade D) of the target lesion by angiographic core lab
Time Frame: Peri-Procedural
Measure: Number; unit: lesions
Arm/Group | Single-arm
Number analyzed (Participants) | 35
lesions
  Technical Success | 35
  Freedom from Any Serious Flow-Limiting Dissection (D-F) | 35
  Residual Stenosis of less than or equal to 50% | 35
Statistical Analysis 1: Comparison: Single-arm; Test type: Other — The primary effectiveness hypothesis is: H0: ΠE ≤ PGE vs. HA: ΠE > PGE, where ΠE is the proportion of target lesions with technical success and PG is the effectiveness Performance Goal. One-sided statistical significance level of 0.025 = α. The hypothesis will be tested using a one-sided Exact Binomial Test; p < .025, Fisher Exact

3. Secondary Outcome: Serious Angiographic Complications
Description: Defined as flow-limiting dissection (≥ Grade D), perforation, distal embolization, or acute vessel closure as assessed by the angiographic core laboratory.
Time Frame: Peri-Procedural
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Single-arm
Number analyzed (Participants) | 35
Number analyzed (Lesions) | 35
Lesions | 0

4. Secondary Outcome: IVL Technical Success (Post- Dilatation)
Description: Defined as post-dilatation residual stenosis ≤50% without flow-limiting dissection (≥ Grade D) of the target lesion, assessed by angiographic core laboratory (measured immediately following mandatory post-dilatation).
Time Frame: Peri-Procedural
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Single-arm
Number analyzed (Participants) | 35
Number analyzed (Lesions) | 35
Lesions
  IVL Technical Success (Post-dilatation) | 30
  Freedom from Any Serious Flow-Limiting Dissection (D-F) | 34
  Residual Stenosis ≤ 50% | 31

5. Secondary Outcome: IVL Device Success
Description: Defined as the ability to deliver, advance across the target lesion, pressurize, pulse, flush, and retrieve the Javelin IVL Catheter
Time Frame: Peri-Procedural
Measure: Number; unit: Javelin Catheters
Units Other Than Participants: Javelin Catheters
Arm/Group | Single-arm
Number analyzed (Participants) | 35
Number analyzed (Javelin Catheters) | 44
Javelin Catheters | 41

6. Secondary Outcome: Technical Success (Final)
Description: Defined as final residual stenosis of ≤30% without flow-limiting dissection (≥ Grade D) of the target lesion by angiographic core laboratory
Time Frame: Peri-Procedural
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Single-arm
Number analyzed (Participants) | 35
Number analyzed (lesions) | 35
lesions
  IVL Technical Success (Final) | 25
  Freedom from Any Serious Flow-Limiting Dissection (D-F) | 35
  Residual Stenosis ≤ 30% | 25

7. Secondary Outcome: MAEs at 6-months Post Procedure
Description: Major Adverse Events (MAEs) at 6 months defined as a composite of:
  * Cardiovascular Death
  * Clinically-driven Target Lesion Revascularization
  * Unplanned Target Limb Amputation (Above the Ankle)
Time Frame: 6 Months Post-Procedure
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: MAEs at 12-months Post Procedure
Description: Major Adverse Events (MAEs) at 12 months defined as a composite of:
  * Cardiovascular Death
  * Clinically-driven Target Lesion Revascularization
  * Unplanned Target Limb Amputation (Above the Ankle)
Time Frame: 12 Months Post-Procedure
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Primary Patency at 12-Months
Description: * Above the knee lesions: freedom from ≥50% restenosis as determined by Duplex Ultrasound (DUS) and freedom from Clinically-Driven Target Lesion Revascularization (CD-TLR)
  * Below the knee lesions: freedom from both total occlusion (100% diameter stenosis by DUS) in all of the target lesions in a flow pathway, as well as a CD-TLR
Time Frame: 12-Months Post Procedure
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 30-Days
Arm/Group | Single-arm
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 8/35
Other Adverse Events (participants affected / at risk) | 17/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm (N=35)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complications (Injury, poisoning and procedural complications) | 2 (2)
Toe amputation (Surgical and medical procedures) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral artery restenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm (N=35)
Vascular procedure complications (Injury, poisoning and procedural complications) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Toe amputation (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT05058456/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT05058456/SAP_001.pdf